CLINICAL TRIAL: NCT03434002
Title: Virtual Reality Simulation for Teaching and Assessment of Anesthesia Crisis Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 15-9985
Record Dates: First submitted 2018-01-17; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Patient Simulation
Keywords: Virtual Reality Simulation; Teaching and Assessment; Anesthesia Crisis Management

STUDY DESIGN:
Intervention Model Description: 1. building the technical components for interaction within the virtual reality environment (phase 1);
  2. application of this virtual reality in medical training (phase 2) and
  3. measurement of training effectiveness with this Virtual Reality simulator against mannequin based training (phase 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): Randomized 15 residents out of 30 Post Graduate Year 1 or 2 anesthesia residents (not involved in initial Virtual Reality testing) will be receive Local Anesthetic Systemic Toxicity simulation training by Virtual Reality simulation
  Interventions: Other: Training by Virtual Reality Simulation
- Arm-B (Experimental): Randomized other 15 residents out of 30 Post Graduate Year 1 or 2 anesthesia residents (not involved in initial Virtual Reality testing) will be receive Local Anesthetic Systemic Toxicity simulation training by mannequin based simulation
  Interventions: Other: Training by Mannequin Based Simulation

INTERVENTIONS:
Other: Training by Virtual Reality Simulation — Those Randomized 15 residents will be receive Local Anesthetic Systemic Toxicity simulation training by Virtual Reality simulation and after two weeks, they will be evaluated by investigators by using the same performance evaluation tool.
  Arms: Arm-A
Other: Training by Mannequin Based Simulation — Randomized other 15 residents will be receive Local Anesthetic Systemic Toxicity simulation training by mannequin based simulation and after two weeks, they will be evaluated by investigators by using the same performance evaluation tool.
  Arms: Arm-B

SUMMARY:
In this study, Investigators are going to develop and test a device to apply virtual reality simulation to improve and help for teaching and assessment of anesthesia crisis management.

DETAILED DESCRIPTION:
Competency based medical education (CBME) is an outcomes-based approach to the design, implementation, assessment, and evaluation of medical education. The goals of Competency Based Medical Education are to improve patient safety, patient health outcomes, and enhance the competence and performance of individuals, groups and teams. Simulation-based training is a proven effective method to improve the skills and competency of the student by permit-ting repetitive practice before an actual procedure is performed on real patients.

e Virtual reality simulation has been used successfully to teach technical skills such as laparoscopic surgery, carotid stenting, gall bladder surgery, and knee arthroscopy.

The specific aims of this project are:

1. Build a multi-user, multi-site virtual reality simulator for anesthesia management and team training
2. Evaluate the simulation as a tool for competency based medical education
3. Compare the effectiveness of the simulator with mannequin based simulator for competency based medical education.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia resident or fellow volunteers from University of Toronto

Exclusion Criteria:

* Unwilling to enter the study
* Previous experience with simulator based teaching on local anesthetic systemic toxicity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of tasks correctly performed | 1 hour
  The primary outcome in performance evaluation is the number of tasks correctly performed during management of the Local Anesthetic Systemic Toxicity event. Investigators will use the same performance evaluation tool.
  The performance evaluation tool will assess the trainee's performance (i.e., medical management of Local Anesthetic Systemic Toxicity) per performance evaluation tool

SECONDARY OUTCOMES:
use the Anesthesiologists' Non-Technical Skills (ANTS) tool | 1 hour
  The Investigators will use the anesthesiologists' non-technical skills (ANTS) tool in the Local Anesthetic Systemic Toxicity Event (Data Collection Tools, Supplemental Digital Content 2, http://links.lww.com/AAP/A45) as described by Neal.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, Principal Investigator — Toronto Western Hospital, University Health Network, University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACGME Outcome Project: Table of Toolbox Methods. (Accessed 1 Sept 2015, at http://njms.rutgers.edu/culweb/medical/documents/ToolboxofAssessmentMethods.pdf).
- [Result] McGaghie WC, Issenberg SB, Petrusa ER, Scalese RJ. A critical review of simulation-based medical education research: 2003-2009. Med Educ. 2010 Jan;44(1):50-63. doi: 10.1111/j.1365-2923.2009.03547.x. PMID 20078756
- [Result] Salas E, DiazGranados D, Weaver SJ, King H. Does team training work? Principles for health care. Acad Emerg Med. 2008 Nov;15(11):1002-9. doi: 10.1111/j.1553-2712.2008.00254.x. Epub 2008 Oct 1. PMID 18828828
- [Result] Sorbero ME, Farley DO, Mattke S, Lovejoy S. Outcome measures for effective teamwork in inpatient care (RAND technical report TR-462-AHRQ). Arlington, VA: RAND Corporation, 2008.
- [Result] Ziv A, Ben-David S, Ziv M. Simulation based medical education: an opportunity to learn from errors. Med Teach. 2005 May;27(3):193-9. doi: 10.1080/01421590500126718. PMID 16011941
- [Result] Alonso A, Baker DP, Holtzman A, et al. Reducing medical error in the military health system: How can team training help? Hum Resour Manag Rev. 2006;16:396-415.
- [Result] Leblanc VR. Review article: simulation in anesthesia: state of the science and looking forward. Can J Anaesth. 2012 Feb;59(2):193-202. doi: 10.1007/s12630-011-9638-8. Epub 2011 Dec 17. PMID 22179792
- [Result] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Result] Grantcharov TP, Kristiansen VB, Bendix J, Bardram L, Rosenberg J, Funch-Jensen P. Randomized clinical trial of virtual reality simulation for laparoscopic skills training. Br J Surg. 2004 Feb;91(2):146-50. doi: 10.1002/bjs.4407. PMID 14760660
- [Result] Nguyen N, Elliott JO, Watson WD, Dominguez E. Simulation Improves Nontechnical Skills Performance of Residents During the Perioperative and Intraoperative Phases of Surgery. J Surg Educ. 2015 Sep-Oct;72(5):957-63. doi: 10.1016/j.jsurg.2015.03.005. Epub 2015 Apr 21. PMID 25911460
- [Result] Neal JM, Hsiung RL, Mulroy MF, Halpern BB, Dragnich AD, Slee AE. ASRA checklist improves trainee performance during a simulated episode of local anesthetic systemic toxicity. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):8-15. doi: 10.1097/AAP.0b013e31823d825a. PMID 22157743
- [Result] Koutantji, Maria, et al.